CLINICAL TRIAL: NCT02513810
Title: A Randomized Controlled Comparison Between One Versus More Than Six Months of Dual Antiplatelet Therapy After Biolimus A9-eluting Stent Implantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2015-0040
Record Dates: First submitted 2015-07-31; First posted 2015-08-03 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Short-term DAPT after Biofreedom (Experimental)
  Interventions: Device: BioFreedom with 1 month DAPT
- Long-term DAPT after BioMatrix or Ultimaster (Active Comparator)
  Interventions: Device: BioMatrix or Ultimaster with 6 to 12 months DAPT

INTERVENTIONS:
Device: BioFreedom with 1 month DAPT — The cath lab will follow site standard operating procedures for PTCA and stenting. Information will be collected and recorded on the treated study vessel including angiographic parameters. Dual antiplatelet therapy after PCI will be continued for 1 month.
  Arms: Short-term DAPT after Biofreedom
Device: BioMatrix or Ultimaster with 6 to 12 months DAPT — The cath lab will follow site standard operating procedures for PTCA and stenting. Information will be collected and recorded on the treated study vessel including angiographic parameters. Dual antiplatelet therapy after PCI will be the duration of dual antiplatelet therapy will be 6 to 12 months at the discretion of the interventionist.
  Arms: Long-term DAPT after BioMatrix or Ultimaster

SUMMARY:
DES are preferred over BMS for most patients, however prolonged dual antiplatelet therapy is required for patients treated with DES for prevention of late or very late stent thrombosis. which increases a risk of major bleeding. BioFreedom is a Biolimus A9-coated stent that consists of a stainless steel stent platform with a textured abluminal surface without use of any polymer in the coating. Biolimus A9 rapid release and polymer-free property may give BioFreedom the advantages of both DES and BMS that may require less duration of DAPT. BioMatrix Flex, Biolimus-eluting stent with biodegradable polymer, also demonstrated safety and efficacy. We will compare these two difference types of Biolimus A9-eluting stents with different duration of DAPT. With proven adequate and safe duration, we will compare between one versus more than six months of dual antiplatelet therapy after Biolimus A9-eluting stents implantation using different properties of BioFreedom and BioMatrix Flex.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 19 years old
* Patients with ischemic heart disease who are considered for coronary revascularization with PCI
* Significant coronary de novo lesion

Exclusion Criteria:

* Acute myocardial infarction
* Complex lesion morphologies such as aorta-ostial, unprotected left main, chronic total occlusion, graft, thrombosis, heavy calcified (definite calcified lesions on angiogram) or extremely tortuous lesion
* Need to use of dual antiplatelet therapy more than 1 month because of other medical conditions
* Cardiogenic shock or experience of cardiopulmonary resuscitation
* Contraindication or hypersensitivity to Biolimus A9, stainless steel, heparin, antiplatelet agents or contrast media
* History of documented prior cerebrovascular attack within 6 months
* Treated with any stent within 3 months
* Reference vessel diameter <2.25 mm or >4.0 mm
* Pregnant women or women with potential childbearing
* Inability to follow the patient over the period of 1 year after enrollment, as assessed by the investigator
* Inability to understand or read the informed content

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3020 (Estimated)
Dates: Start 2015-12-02 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Composite of major adverse cardiovascular events | 1 year
  events including cardiac death, nonfatal myocardial infarction, target vessel revascularization, major bleeding and cerebrovascular accident

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Jin IT, Kim Y, Heo SJ, Lee YJ, Lee SJ, Hong SJ, Ahn CM, Kim JS, Cho DK, Ko YG, Choi D, Hong MK, Kim BK. Comparison of Short-term and Standard Duration Dual Antiplatelet Therapy in Elderly Patients: A Pooled Analysis of Five Korean Randomized Clinical Trials. Korean Circ J. 2025 Dec;55(12):1125-1137. doi: 10.4070/kcj.2025.0093. Epub 2025 Jul 14. PMID 41044734
- [Derived] Lee YJ, Cho JY, Yun KH, Lee SJ, Hong SJ, Ahn CM, Kim BK, Ko YG, Choi D, Hong MK, Jang Y, Kim JS. Impact of one-month DAPT followed by aspirin monotherapy in patients undergoing percutaneous coronary intervention according to clinical presentation: a post hoc analysis of the randomised One-Month DAPT trial. EuroIntervention. 2022 Aug 19;18(6):471-481. doi: 10.4244/EIJ-D-22-00135. PMID 35470799
- [Derived] Hong SJ, Kim JS, Hong SJ, Lim DS, Lee SY, Yun KH, Park JK, Kang WC, Kim YH, Yoon HJ, Won H, Nam CM, Ahn CM, Kim BK, Ko YG, Choi D, Jang Y, Hong MK; One-Month DAPT Investigators. 1-Month Dual-Antiplatelet Therapy Followed by Aspirin Monotherapy After Polymer-Free Drug-Coated Stent Implantation: One-Month DAPT Trial. JACC Cardiovasc Interv. 2021 Aug 23;14(16):1801-1811. doi: 10.1016/j.jcin.2021.06.003. Epub 2021 Jul 28. PMID 34332946